CLINICAL TRIAL: NCT01206738
Title: Developing and Evaluating Interventions to Reduce Inappropriate Prescribing by General Practitioners of Antibiotics for Upper Respiratory Tract Infections: an RCT to Compare Paper-based and Web-based Modelling Experiments
Brief Title: Developing and Evaluating Interventions to Reduce Inappropriate Prescribing of Antibiotics in Primary Care
Acronym: WIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: University of Aberdeen (Other); Newcastle University (Other); University of Southampton (Other); Chief Scientist Office of the Scottish Government (Other Government); Scottish Primary Care Research Network (Unknown); Scottish School of Primary Care (Unknown)
Responsible Party: Principal Investigator, Shaun Treweek, Senior Lecturer, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2010PS10; CZH/4/610 (Other Grant/Funding Number: Chief Scientist Office)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Antibiotic Prescribing by GPs for URTI

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Persuasive communication (Experimental): The persuasive intervention aimed to reinforce the GP's beliefs about the positive consequences of managing sore throat without prescribing antibiotics.
  Interventions: Behavioral: Persuasive communication
- Alternative intervention (Experimental): This intervention was an action plan, supporting the GP to deal with two difficult prescribing situations: 1) a distressed patient (or often distressed parent of a child patient) 2) a patient demanding an antibiotic
  Interventions: Behavioral: Action plan
- General information (Active Comparator): No additional information was provided; the general information was the information already available to GPs about antibiotic prescribing.
  Interventions: Behavioral: General intervention

INTERVENTIONS:
Behavioral: Persuasive communication — The persuasive intervention aimed to reinforce the GP's beliefs about the positive consequences of managing sore throat without prescribing antibiotics.
  Arms: Persuasive communication
Behavioral: Action plan — This intervention was an action plan, supporting the GP to deal with two difficult prescribing situations: 1) a distressed patient (or often distressed parent of a child patient) 2) a patient demanding an antibiotic
  Arms: Alternative intervention
Behavioral: General intervention — No additional information was provided; the general information was the information already available to GPs about antibiotic prescribing.
  Arms: General information

SUMMARY:
1. Do paper-based and web-based intervention modelling experiments (the methodology we are developing) identify the same predictors of GP behaviour regarding prescribing of antibiotics for upper respiratory tract infections?
2. Can a web-based IME system provide trialists with richer and more predictive information upon which to base the development of behavioural change interventions than paper-based IME systems?

DETAILED DESCRIPTION:
The NHS needs effective quality improvement interventions to be put into clinical practice, which requires effective behaviour change interventions. Intervention modelling experiments (IMEs) are a way of exploring and refining an intervention before moving to a full-scale trial. They do this by delivering key elements of the intervention in a simulation that approximates clinical practice by, for example, presenting GPs with a clinical scenario about making a treatment decision. Earlier IMEs have been paper-based, which limits what can be done in the simulation.

Web-based IMEs provide the potential for better clinical simulations, which have the potential to lead to better interventions. The current proposal will run a full, web-based IME involving 250 GPs that will advance the methodology of IMEs by directly comparing results with an earlier paper-based IME. Moreover, the web-based IME will evaluate an intervention that can be put into a full-scale trial that aims to reduce antibiotic prescribing in primary care. Reducing inappropriate prescribing of antibiotics in general practice is a national priority; indeed, antibiotic use is increasing in the UK and Scotland's prescribing is second highest amongst UK administrations. More effective behaviour change interventions are needed and this proposal will develop one such intervention and a system to model and test future interventions. This system will be applicable to any situation in the NHS where behaviour needs to be modified, including interventions aimed directly at the public.

ELIGIBILITY:
Inclusion Criteria:

* GPs in Scotland.

Exclusion Criteria:

* Unable to obtain both an email address and a postal address for the GP.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Treweek, PhD, Principal Investigator — University of Dundee
Locations (1):
- University of Dundee, Dundee, Tayside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are no patient-level data in this trial because no patients were involved. More information about the study and what was collected can be obtained from the Shaun Treweek at streweek@mac.com.

REFERENCES:
- [Background] Treweek S, Ricketts IW, Francis J, Eccles M, Bonetti D, Pitts NB, Maclennan G, Sullivan F, Jones C, Weal M, Barnett K. Developing and evaluating interventions to reduce inappropriate prescribing by general practitioners of antibiotics for upper respiratory tract infections: a randomised controlled trial to compare paper-based and web-based modelling experiments. Implement Sci. 2011 Mar 3;6:16. doi: 10.1186/1748-5908-6-16. PMID 21371323
- [Result] Treweek S, Barnett K, Maclennan G, Bonetti D, Eccles MP, Francis JJ, Jones C, Pitts NB, Ricketts IW, Weal M, Sullivan F. E-mail invitations to general practitioners were as effective as postal invitations and were more efficient. J Clin Epidemiol. 2012 Jul;65(7):793-7. doi: 10.1016/j.jclinepi.2011.11.010. Epub 2012 Feb 4. PMID 22306007
- [Result] Treweek S, Bonetti D, Maclennan G, Barnett K, Eccles MP, Jones C, Pitts NB, Ricketts IW, Sullivan F, Weal M, Francis JJ. Paper-based and web-based intervention modeling experiments identified the same predictors of general practitioners' antibiotic-prescribing behavior. J Clin Epidemiol. 2014 Mar;67(3):296-304. doi: 10.1016/j.jclinepi.2013.09.015. Epub 2013 Dec 31. PMID 24388292
- [Result] Treweek S, Francis JJ, Bonetti D, Barnett K, Eccles MP, Hudson J, Jones C, Pitts NB, Ricketts IW, Sullivan F, Weal M, MacLennan G. A primary care Web-based Intervention Modeling Experiment replicated behavior changes seen in earlier paper-based experiment. J Clin Epidemiol. 2016 Dec;80:116-122. doi: 10.1016/j.jclinepi.2016.07.008. Epub 2016 Jul 26. PMID 27470610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For email vs postal study, 880 physicians received email and 880 received postal invitations. 138 and 132 responded respectively. Other recruitment data presented below are for the main trial component, which involved a subset of the 270 (ie. 138+132) responding to the initial invitation.
  See arm descriptions for further explanation.
Pre-assignment Details: Note this study has two parts: 1) an email vs postal invitation study (with 270 enrolled) and 2) a trial involving a subset (172) of those involved in the email vs postal invitation study. The trial enrolled 198 participants in total, with 26 participants not being involved in the email study.
  See arm descriptions for further explanations.
Groups:
- Persuasive Communication: The persuasive intervention aimed to reinforce the GP's beliefs about the positive consequences of managing sore throat without prescribing antibiotics.
  Note: for the Overall study, the best 25% of prescribers completing the email vs postal invitation sub study (which 270 individuals completed) were not eligible by definition (we only wanted to trial our interventions with doctors not prescribing according to best practice). Of the 270, only 201 were eligible. All were invited to participate, along with 313 other family doctors who had not taken part in the email vs. postal invitation study. Of the 514 (201 + 313) invited to the Overall study, 198 responded and these are the participants for the Overall study.
- Alternative Intervention: Action Plan. The work linking simulated prescribing behaviour to predictors of that behaviour suggested that an action plan, detailing situations where GPs found it difficult to not prescribe an antibiotic and offering ways in which the GP could avoid prescribing an antibiotic when this was not necessary.
  Note: for the Overall study, the best 25% of prescribers completing the email vs postal invitation sub study (which 270 individuals completed) were not eligible by definition (we only wanted to trial our interventions with doctors not prescribing according to best practice). Of the 270, only 201 were eligible. All were invited to participate, along with 313 other family doctors who had not taken part in the email vs. postal invitation study. Of the 514 (201 + 313) invited to the Overall study, 198 responded and these are the participants for the Overall study.
- General Information: No information beyond the information that GPs already have from guidelines and other diverse sources (ie. usual care).
  Note: for the Overall study, the best 25% of prescribers completing the email vs postal invitation sub study (which 270 individuals completed) were not eligible by definition (we only wanted to trial our interventions with doctors not prescribing according to best practice). Of the 270, only 201 were eligible. All were invited to participate, along with 313 other family doctors who had not taken part in the email vs. postal invitation study. Of the 514 (201 + 313) invited to the Overall study, 198 responded and these are the participants for the Overall study.
Period: Overall Study
Arm/Group | Persuasive Communication | Alternative Intervention | General Information
Started | 63 | 74 | 61
Completed | 40 | 49 | 42
Not Completed | 23 | 25 | 19

BASELINE CHARACTERISTICS:
Population: GPs across Scotland
Groups:
- Alternative Intervention: Action Plan. The work linking simulated prescribing behaviour to predictors of that behaviour suggested that an action plan, detailing situations where GPs found it difficult to not prescribe an antibiotic and offering ways in which the GP could avoid prescribing an antibiotic when this was not necessary.
- General Information: No information beyond the information that GPs already have from guidelines and other diverse sources (ie. usual care)
- Total: Total of all reporting groups
Arm/Group | Persuasive Communication | Alternative Intervention | General Information | Total
Number analyzed (Participants) | 63 | 74 | 61 | 198
Age, Customized [Mean (Standard Deviation); unit: years] — Age was not collected; we collected years a GP had been qualified
  years
    Years qualified | 22 (9) | 20 (9) | 22 (8) | 21 (9)
Sex/Gender, Customized [Number; unit: participants] — Some participants chose not to respond to the gender question.
  participants
    Female | 27 | 34 | 27 | 88
    Male | 35 | 36 | 32 | 103
Region of Enrollment [Number; unit: participants]
  United Kingdom | 63 | 74 | 61 | 198

OUTCOME MEASURES:

1. Primary Outcome: Number of Simulated Scenarios Where an Antibiotic Was Not Prescribed
Description: Eight simulated clinical scenarios where presented to the GP and he/she was asked whether an antibiotic should be prescribed. The outcome measures was the number of scenarios where an antibiotic was not prescribed.
Time Frame: Immediately after completion of questionnaire
Measure: Mean (Standard Deviation); unit: scenarios
Arm/Group | Persuasive Communication | Alternative Intervention | General Information
Number analyzed (Participants) | 40 | 49 | 42
scenarios | 5 (1.4) | 5 (1.6) | 4.2 (1.1)

2. Primary Outcome: Email vs Postal Recruitment: Number of GPs Completing the First Questionnaire
Description: GPs were randomly allocated to receive their invitation to take part by email or by post. Outcome measure was proportion of GPs responding by completing the first questionnaire
Time Frame: 27/1/20111 - 15/5/2011
Population: 880 physicians received email and 880 received postal invitations. 138 and 132 responded respectively.
Measure: Number; unit: participants
Groups:
- Email: GPs receiving an email invitation
- Post: GPs receiving a postal invitation
Arm/Group | Email | Post
Number analyzed (Participants) | 880 | 880
participants | 138 | 132

ADVERSE EVENTS:
Description: The study was a web-based questionnaire study asking family doctors questions linked to text-based simulated clinical scenarios. This was considered as zero-risk and no adverse event data were recorded and no adverse events were reported by participants.
Arm/Group | Persuasive Communication | Alternative Intervention | General Information
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No